CLINICAL TRIAL: NCT00675220
Title: A Prospective, Open-Labelled, Non-Controlled, Observational Study to Assess the Efficacy and Safety of NovoRapid™ FlexPen™ in the Treatment of Acute Hyperglycemia: A Post-Marketing Surveillance Study
Brief Title: Observational Study to Assess the Efficacy and Safety of NovoRapid™ Flexpen™
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: ANA-1884
Record Dates: First submitted 2008-05-06; First posted 2008-05-09 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Delivery Systems
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Aspart

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: insulin aspart — Start dose and frequency to be prescribed by the physician as a result of the normal clinical evaluation

SUMMARY:
This study is conducted in Asia. The aim of this observational study is to collect efficacy and safety data in diabetic patients with acute hyperglycemia using NovoRapid™ FlexPen™ as per normal clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes mellitus (according to product labelling)

Exclusion Criteria:

* Hypoglycaemia
* Hypersensitivity to insulin aspart or to any of the excipients (according to product labelling)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Diabetes
Sampling Method: Non-Probability Sample
Enrollment: 373 (Actual)
Dates: Start 2007-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Safety profile of Insulin Aspart among Filipino patients | 1-month follow-up for outpatients; 1 month or upon discharge for inpatients whichever comes first

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Manila, Philippines

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com